CLINICAL TRIAL: NCT05933135
Title: Influence of Factor XIII Activity on the Outcome of Gastrointestinal Bleedings
Brief Title: Factor XIII Activity in Gastrointestinal Bleedings
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EK 33-123 ex 20/21
Record Dates: First submitted 2023-02-20; First posted 2023-07-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Factor XIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal factor XIII acitivity: Patients with GI bleeding and normal factor XIII activity
- Reduced factor XIII activity: Patients with GI bleeding and reduced factor XIII activity
  Interventions: Drug: Factor XIII Injection

INTERVENTIONS:
Drug: Factor XIII Injection — Patients could have had an Factor XIII Injection in clinical routine
  Groups: Reduced factor XIII activity

SUMMARY:
The aim of this retrospective study is to investigate the relationship between factor XIII activity and the outcome of gastrointestinal bleedings. Since factor XIII is of great importance in haemostasis and plays a key role in stabilizing the fibrin clot, it can be assumed that a deficiency of factor XIII leads to an unfavorable course of gastrointestinal bleedings. Our hypothesis is that early detection of such a deficiency can prevent a more severe course and that substitution of factor XIII contributes to faster cessation of bleeding, improves patient outcome and reduces the number of red cell concentrates required.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Confirmed diagnosis of gastrointestinal bleeding
* Assessment of factor XIII activity during the gastrointestinal bleeding episode

Exclusion Criteria:

* Age under 18 years
* Diagnosis of hemophilia A or B or other congenital coagulation disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were retrospectively recruited if they suffered an episode of a gastrointestinal bleeding and factor XIII was measured.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Red cell concentrates | 1 year
  Number of red cell concentrates transfused during the hospital stay caused by the gastrointestinal bleeding episode

SECONDARY OUTCOMES:
Hospitalization | 1 year
  Length of the hospital stay caused by the gastrointestinal bleeding episode
Interventions | 1 year
  Number of endoscopic, radiological, and surgical interventions for bleeding treatment within the hospital stay caused by the gastrointestinal bleeding episode
Mortality | 1 year
  In hospital-mortality during the hospital stay caused by the gastrointestinal bleeding episode

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hoegenauer, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No